CLINICAL TRIAL: NCT05816603
Title: Home-based Post-stroke Fatigue Treatment Using Transcranial Direct Current Stimulation (tDCS)
Brief Title: Transcranial Direct Current Stimulation for Post-stroke Fatigue
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-11025409
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Fatigue; Stroke Rehabilitaion
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Real tDCS stimulation (Experimental): Subjects randomized to receive real/active electrical stimulation.
  Interventions: Device: Real Soterix Mini-CT tDCS stimulator
- Sham tDCS stimulation (Sham Comparator): Subjects randomized to receive sham/non-activating electrical stimulation.
  Interventions: Device: Sham Soterix Mini-CT tDCS stimulator

INTERVENTIONS:
Device: Real Soterix Mini-CT tDCS stimulator — Real transcranial electrical stimulation at 2mA intensity will be delivered to the left dorsolateral prefrontal cortex, 20 minutes/day, 14-day duration.
  Arms: Real tDCS stimulation
Device: Sham Soterix Mini-CT tDCS stimulator — Sham stimulation to the left dorsolateral prefrontal cortex, 20 minutes/day, 14-day duration. The device will ramp up and ramp down current delivery from 0 mA -2 mA - 0 mA over 30 seconds at the start of the 20-minute protocol with no active stimulation until the end of the 20 minutes, at which time the 30-second ramp up/ramp down will be repeated.
  Arms: Sham tDCS stimulation

SUMMARY:
The investigators hypothesize that delivery of anodal tDCS to the left frontal head region will reduce fatigue severity following stroke.

DETAILED DESCRIPTION:
The purpose of this study is to investigate transcranial direct current stimulation (tDCS) as a home-based non-pharmacologic intervention for post-stroke fatigue (PSF). Investigators will perform a double-blind, sham-controlled, randomized clinical trial with 24 subjects; 12 will receive sham stimulation and 12 will receive real stimulation. After a baseline assessment, the tDCS device will be applied for 20 minutes, once daily over the left dorsolateral prefrontal cortex (DLPFC), for a total of two weeks. Follow-up assessments with outcome metrics will be completed after the seventh and fourteenth sessions, and one-month following the start date (2 weeks post-treatment). Neuroimaging will be completed at baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >18 years
* Greater than 3 months from first hemorrhagic or ischemic stroke (subacute to chronic), confirmed through neuroimaging (CT or MRI).
* Fatigue severity score average >4 (severe fatigue)
* Willingness to remain stable on pharmacologic therapy through the duration of the study.
* Availability of a caregiver, family member, or friend to be present during the administration of the tDCS intervention.

Exclusion Criteria:

* Metal in the head (except mouth) or implanted cranial or thoracic devices (i.e. pacemaker, DBS stimulator)
* History of seizure
* History of moderate to severe traumatic brain injury
* A score of 10 or more on the PHQ-9 or GAD-7 scale, suggestive of moderate to severe depression/anxiety.
* A score of less than 21 on the MoCA suggesting major neurocognitive disorder.
* Signs of skin rash, infection, or laceration in the supraorbital region where the tDCS will be applied.
* Inability to provide informed consent
* Other major neurological, medical, or psychiatric illnesses that could confound results in the opinion of the site investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline Fatigue Severity Scale - 7 (FSS-7) | Screening (-1 to -14 days), Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52))
  Fatigue Severity. This seven item scale measures fatigue severity and it's effect on a person's lifestyle and activities. Items are scored on a seven point scale. Minimum score = 7, maximum score = 49 with higher score indicating greater fatigue severity.

SECONDARY OUTCOMES:
Mean change from baseline Stroke Specific Quality Of Life scale (SS-QOL) | Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Quality of Life. Assesses health related quality of life, specific to individuals with stroke. Composed of 49 items, score on a 5 point guttman type scale. Scores range from 49 to 245, with higher score indicating better functioning.
Mean change from baseline Patient Health Questionnaire - 9 (PHQ-9) | Screening (-1 to -14 days), Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Depression. A multipurpose instrument for screening, measuring, and monitoring severity of depression. Scores range from 0-27, with higher score indicating greater severity of depression.
Mean change from baseline Generalized Anxiety Disorder - 7 (GAD-7) | Screening (-1 to -14 days), Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Anxiety. A multipurpose instrument for screening, measuring, and monitoring severity of anxiety. Scores range from 0-21, with higher score indicating greater severity of anxiety.
Mean change from baseline PROMIS-sleep disturbance | Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Sleep. A domain focused self report of global, physical, mental, and social health for those living with a chronic condition. Computer adapted test with higher scores indicating more sleep disturbance. Results reported as a T-score with range from 10-90 based on the United States general population average score of 50 and standard deviation of 10. Higher t-score indicates greater sleep disturbance.
Mean change from baseline Symbol Digit Modalities Test (SDMT) | Baseline (Day 1), Post-Treatment (Day 14-21)
  Cognition. A measure of cognitive processing speed and attention. Scores range from 0-120, with higher scores better performance.
Mean change from baseline Test of Variables of Attention (T.O.V.A) | Baseline (Day 1), Post-Treatment (Day 14-21)
  Cognition. A computerized test that measures short-term memory, with scores from 85-115 indicating a normal result. Response time, response time variability, commissions, and omissions are also recorded. A higher total number correct score indicates better performance.
Mean change from baseline Montreal cognitive assessment (MoCA) | Baseline (Day 1), Post-Treatment (Day 14-21)
  Cognition. A brief screening tool to assess global cognitive functioning and detect mild cognitive dysfunction. Scored from 0-30 with higher score indicating better performance.
Mean Client Satisfaction Questionnaire - 8 (CSQ-8) | During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Feasibility. This tool is a self-report measure participant satisfaction with the intervention. Scored 8-32 with higher scores indicating greater satisfaction.
Mean change from baseline Frenchay activities index | Baseline (Day 1), During-treatment (Day 7-9), Post-Treatment (Day 14-21), 1 Month Post-Treatment (Day 45-52)
  Activities of Daily Living (ADLs). A measure of instrumental ADLs (domestic chores, leisure/work, outdoor activities) for individuals recovering from stroke. Scored from 15-60 with higher score indicating improved functioning.
Change in resting state brain functional connectivity. | Baseline (Day 1), Post-treatment (Day 14-21)
  Change in functional connectivity in the active vs. the sham arms assessed by a resting state functional magnetic resonance imaging scan (rs-fMRI).

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Stilling, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, 525 E. 68th St, Baker Pavilion, F-2106, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: To achieve aims in the approved proposal. Proposals may be submitted to the study P.I. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years following publication.